CLINICAL TRIAL: NCT00378352
Title: Effects of Erythropoietin on Infarct Size and Left Ventricular Remodeling in Survivors of Large Myocardial Infarctions
Brief Title: REVEAL: Reduction of Infarct Expansion and Ventricular Remodeling With Erythropoietin After Large Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 999905255; 05-AG-N255 (Other: NIH)
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Acute ST Elevation Myocardial Infarction
Keywords: Acute Myocardial Infarction; Left Ventricular Remodeling; Cardiac Magnetic Resonance Imaging; Endothelial Progenitor Cells; Infarct Size
MeSH Terms: conditions — Ventricular Remodeling | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose Escalation Safety (Placebo Comparator): The objective of the first phase is to evaluate the safety of escalating doses of Epoetin alfa in patients with STEMIs.
  Interventions: Drug: Epoetin alfa
- Single Dose Efficacy (Placebo Comparator): Single parenteral administration of 60000 U of epoetin alfa. The objectives of the second phase are to investigate the effects of the highest safe dose on infarct size, left ventricular remodeling and endothelial progenitor cells.
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: Epoetin alfa — Randomized
  Other Names: PROCRIT

SUMMARY:
The purpose of this study is to evaluate whether erythropoietin can help limit the damage to the heart in patients with acute heart attacks.

DETAILED DESCRIPTION:
REVEAL is a randomized, double-blinded, placebo-controlled, parallel phase II clinical study that will evaluate the effects of erythropoietin administration on infarct size, left ventricular remodeling and circulating endothelial progenitor cells in patients with large myocardial infarctions (MI). The study will be conducted in two phases: a dose-escalation safety phase and a single dose efficacy phase. Eligible patients who present to the hospital with an acute ST-elevation MI and who agree to participate in this study will be randomly assigned to receive a single infusion of study medication consisting either of erythropoietin or placebo. The size of the infarction and the dimensions of the heart will be assessed by cardiac magnetic resonance imaging (MRI) within 2-6 days of the infusion of the study medication, and again approximately 3 months later.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than 21 years

Acute ST-elevation myocardial infarction

Referral for primary or rescue angioplasty

Revascularization procedure within 8 hours from the onset of ischemic symptoms

TIMI (Thrombolysis in myocardial infarction) flow grade 0 or 1 in the culprit coronary artery at the beginning of coronary angiography

Successful revascularization of infarct-related artery

EXCLUSION CRITERIA:

Clinical indication for erythropoietin

STEMI (ST-elevation myocardial infarction) due to occlusion of a branch vessel

Any history of prior MI, PCI (Percutaneous coronary intervention), CABG (Coronary artery bypass graft), cardiomyopathy, myocarditis, or CHF (congestive heart failure)

Hypersensitivity to human albumin, mammalian cell-derived products, or erythropoietin

Hematocrit greater than 42% in men or greater than 40% in women at the time of study drug administration

Uncontrolled hypertension at the time of study drug administration

Cardiogenic shock

Need for coronary surgical revascularization as determined at the time of the index coronary catheterization

History of hypercoagulable disorder, thromboembolic event, or venous thrombosis

History of stroke or TIA (transient ischemic attack)

History of seizures

Contraindication to MRI

Pregnancy or nursing mother

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2005-09; Primary Completion 2009-07 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward G Lakatta, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (16):
- United States (16):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Miami, School of Medicine, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - New York Methodist Hospital, Brooklyn, New York
  - Cornell University, New York, New York
  - NY Presbyterian Hospital, New York, New York
  - Weill Medical College, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Penn State Heart and Vascular Institute, Hershey, Pennsylvania
  - Nashville Cardiovascular Magnetic Resonance Institute, Brentwood, Tennessee
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogoyevitch MA. An update on the cardiac effects of erythropoietin cardioprotection by erythropoietin and the lessons learnt from studies in neuroprotection. Cardiovasc Res. 2004 Aug 1;63(2):208-16. doi: 10.1016/j.cardiores.2004.03.017. PMID 15249178
- [Background] Parsa CJ, Matsumoto A, Kim J, Riel RU, Pascal LS, Walton GB, Thompson RB, Petrofski JA, Annex BH, Stamler JS, Koch WJ. A novel protective effect of erythropoietin in the infarcted heart. J Clin Invest. 2003 Oct;112(7):999-1007. doi: 10.1172/JCI18200. PMID 14523037
- [Background] Maiese K, Li F, Chong ZZ. New avenues of exploration for erythropoietin. JAMA. 2005 Jan 5;293(1):90-5. doi: 10.1001/jama.293.1.90. PMID 15632341
- [Background] Povsic TJ, Najjar SS, Prather K, Zhou J, Adams SD, Zavodni KL, Kelly F, Melton LG, Hasselblad V, Heitner JF, Raman SV, Barsness GW, Patel MR, Kim RJ, Lakatta EG, Harrington RA, Rao SV. EPC mobilization after erythropoietin treatment in acute ST-elevation myocardial infarction: the REVEAL EPC substudy. J Thromb Thrombolysis. 2013 Nov;36(4):375-83. doi: 10.1007/s11239-013-0944-6. PMID 23700090
- [Result] Najjar SS, Rao SV, Melloni C, Raman SV, Povsic TJ, Melton L, Barsness GW, Prather K, Heitner JF, Kilaru R, Gruberg L, Hasselblad V, Greenbaum AB, Patel M, Kim RJ, Talan M, Ferrucci L, Longo DL, Lakatta EG, Harrington RA; REVEAL Investigators. Intravenous erythropoietin in patients with ST-segment elevation myocardial infarction: REVEAL: a randomized controlled trial. JAMA. 2011 May 11;305(18):1863-72. doi: 10.1001/jama.2011.592. PMID 21558517
- [Derived] Melloni C, Rao SV, Povsic TJ, Melton L, Kim RJ, Kilaru R, Patel MR, Talan M, Ferrucci L, Longo DL, Lakatta EG, Najjar SS, Harrington RA. Design and rationale of the Reduction of Infarct Expansion and Ventricular Remodeling with Erythropoietin after Large Myocardial Infarction (REVEAL) trial. Am Heart J. 2010 Nov;160(5):795-803.e2. doi: 10.1016/j.ahj.2010.09.007. PMID 21095264

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 28 US sites between October 2006 and February 2010 and included 222 patients with STEMI who underwent successful percutaneous coronary intervention (PCI) as a primary or rescue reperfusion strategy
Groups:
- Efficacy Phase 60,000 Units Epoetin Alfa: Prospective, randomized, double-blind, placebo-controlled trial Single dose 60000 U of epoetin alfa
- Efficacy Phase Placebo: Single dose placebo
Period: Dose Escalation 15,000 Units
Arm/Group | Dose Escalation 15,000 Units Epoetin Alfa | Dose Escalation 30,000 Units Epoetin Alfa | Dose Escalation 60,000 Units Epoetin Alfa | Dose Escalation Placebo | Efficacy Phase 60,000 Units Epoetin Alfa | Efficacy Phase Placebo
Started | 20 | 0 | 0 | 11 | 0 | 0
Safety Analysis | 19 | 0 | 0 | 11 | 0 | 0
Completed | 15 | 0 | 0 | 10 | 0 | 0
Not Completed | 5 | 0 | 0 | 1 | 0 | 0
Period: Dose Escalation 30,000 Units
Arm/Group | Dose Escalation 15,000 Units Epoetin Alfa | Dose Escalation 30,000 Units Epoetin Alfa | Dose Escalation 60,000 Units Epoetin Alfa | Dose Escalation Placebo | Efficacy Phase 60,000 Units Epoetin Alfa | Efficacy Phase Placebo
Started | 0 | 19 | 0 | 11 | 0 | 0
Safety Analysis | 0 | 20 (One participant randomized to 60,000 units received 30,000 units) | 0 | 11 | 0 | 0
Completed | 0 | 16 | 0 | 9 | 0 | 0
Not Completed | 0 | 3 | 0 | 2 | 0 | 0
Period: Dose Escalation 60,000 Units
Arm/Group | Dose Escalation 15,000 Units Epoetin Alfa | Dose Escalation 30,000 Units Epoetin Alfa | Dose Escalation 60,000 Units Epoetin Alfa | Dose Escalation Placebo | Efficacy Phase 60,000 Units Epoetin Alfa | Efficacy Phase Placebo
Started | 0 | 0 | 20 | 11 | 0 | 0
Safety Analysis | 0 | 0 | 19 | 11 | 0 | 0
Completed | 0 | 0 | 17 | 10 | 0 | 0
Not Completed | 0 | 0 | 3 | 1 | 0 | 0
Period: Efficacy Phase
Arm/Group | Dose Escalation 15,000 Units Epoetin Alfa | Dose Escalation 30,000 Units Epoetin Alfa | Dose Escalation 60,000 Units Epoetin Alfa | Dose Escalation Placebo | Efficacy Phase 60,000 Units Epoetin Alfa | Efficacy Phase Placebo
Started | 0 | 0 | 0 | 0 | 65 | 66
Safety Analysis | 0 | 0 | 0 | 0 | 67 (Two participants randomized to placebo received 60,000 units Epoetin alfa) | 64
Completed | 0 | 0 | 0 | 0 | 54 | 59
Not Completed | 0 | 0 | 0 | 0 | 11 | 7

BASELINE CHARACTERISTICS:
Population: One participant was not included
Groups:
- Epoetin Alfa; Placebo: Dose escalation and efficacy phases
- Total: Total of all reporting groups
Arm/Group | Epoetin Alfa | Placebo | Total
Number analyzed (Participants) | 123 | 99 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (12.4) | 55.6 (12.5) | 56 (12)
Age, Customized [Count of Participants; unit: Participants]
  Less than 70 years | 103 | 81 | 184
  Greater than or equal to 70 years | 20 | 18 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 100 | 78 | 178
Region of Enrollment [Number; unit: participants]
  United States | 123 | 99 | 222

OUTCOME MEASURES:

1. Primary Outcome: Infarct Size in the Territory of the Infarct Related Artery
Description: Infarct size, expressed as percentage of LV mass, assessed by cardiac magnetic resonance (CMR) imaging.
Time Frame: performed 2 to 6 days after study medication administration (first CMR)
Population: Analysis only performed on subjects who completed the CMR examination
Measure: Mean (Standard Deviation); unit: percentage of LV mass
Groups:
- Epoetin Alfa: Highest dose cohort (60,000 U of epoetin alfa)
- Placebo: Placebo for the highest dose
Arm/Group | Epoetin Alfa | Placebo
Number analyzed (Participants) | 68 | 68
percentage of LV mass | 15.8 (10.3) | 15.0 (10.0)

2. Secondary Outcome: Infarct Size in the Territory of the Infarct Related Artery
Description: Infarct size, expressed as percentage of LV mass, assessed by cardiac magnetic resonance (CMR) imaging.
Time Frame: 12 ± 2 weeks after study medication
Population: Analysis only performed on subjects who completed the CMR examination
Measure: Mean (Standard Deviation); unit: percentage of LV mass
Arm/Group | Epoetin Alfa | Placebo
Number analyzed (Participants) | 61 | 63
percentage of LV mass | 10.6 (8.6) | 10.4 (7.6)

3. Secondary Outcome: LV Ejection Fraction
Time Frame: 2 to 6 days after study medication administration (first CMR) and 12 ± 2 weeks later (second CMR)
Population: Analysis only performed on subjects who completed this component of the CMR examination
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Epoetin Alfa | Placebo
Number analyzed (Participants) | 68 | 70
percent
  First CMR | 48.2 (9.1) | 48.9 (8.7)
  Second CMR: number analyzed (Participants) | 61 | 63
  Second CMR | 52.5 (9.3) | 52.0 (8.8)

4. Secondary Outcome: LV Volume Indexed to BSA
Time Frame: 2 to 6 days after study medication administration (first CMR) and 12 ± 2 weeks later (second CMR)
Population: Analysis only performed on subjects who completed this component of the CMR examination
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Epoetin Alfa | Placebo
Number analyzed (Participants) | 65 | 68
ml/m^2
  End systolic, First CMR | 34.7 (14.7) | 32.6 (10.6)
  End systolic, Second CMR: number analyzed (Participants) | 61 | 62
  End systolic, Second CMR | 34.1 (14.0) | 32.0 (11.7)
  End diastolic, First CMR | 65.6 (18.2) | 63.4 (15.4)
  End diastolic, Second CMR: number analyzed (Participants) | 61 | 62
  End diastolic, Second CMR | 70.0 (17.1) | 66.6 (19.1)

5. Secondary Outcome: LV Mass Indexed to BSA
Time Frame: 2 to 6 days after study medication administration (first CMR) and 12 ± 2 weeks later (second CMR)
Population: Analysis only performed on subjects who completed this component of the CMR examination
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Epoetin Alfa | Placebo
Number analyzed (Participants) | 68 | 69
g/m^2
  First CMR | 74.2 (15.2) | 69.2 (13.0)
  Second CMR: number analyzed (Participants) | 61 | 63
  Second CMR | 67.3 (14.7) | 61.8 (14.1)

6. Secondary Outcome: Vital Signs
Time Frame: baseline, 24 hours, 48 hours, 14 (+/- 5) days, and 30 (+/- 5) days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Epoetin Alfa | Placebo
Number analyzed (Participants) | 125 | 97
mmHg
  SBP, baseline | 129.7 (17.9) | 126.2 (18.7)
  SBP at 24 hours | 118.7 (19.1) | 112.9 (16.7)
  SBP at 48 hours | 114.3 (18.3) | 114.3 (16.3)
  SBP, 14 days | 119.2 (18.9) | 115.2 (14.3)
  SBP, 30 days | 117.4 (16.3) | 117.9 (16.5)
  DBP, baseline | 78.5 (12.7) | 75.8 (13.8)
  DBP, 24 hours | 70.5 (12.9) | 66.3 (11.0)
  DBP, 48 hours | 68.0 (11.5) | 67.9 (11.5)
  DBP, 14 days | 71.2 (10.9) | 69.2 (9.8)
  DBP, 30 days | 71.0 (10.3) | 71.3 (10.8)

7. Secondary Outcome: Hemoglobin Levels
Time Frame: baseline, 24 hours, 48 hours, 14 (+/- 5) days, and 30 (+/- 5) days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa | Placebo
Number analyzed (Participants) | 125 | 97
g/dL
  Baseline | 13.8 (1.4) | 13.6 (1.7)
  24 hours | 13.4 (1.5) | 13.1 (1.7)
  48 hours | 13.3 (1.7) | 13.1 (1.8)
  14 days | 14.1 (1.4) | 13.5 (1.5)
  30 days | 14.2 (1.4) | 13.7 (1.5)

8. Secondary Outcome: Reticulocyte Counts
Time Frame: baseline, 24 hours, 48 hours, 14 (+/- 5) days, and 30 (+/- 5) days
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Epoetin Alfa | Placebo
Number analyzed (Participants) | 125 | 97
percentage of red blood cells
  Baseline | 1.4 (0.5) | 1.3 (0.5)
  24 hours | 1.6 (0.5) | 1.3 (0.6)
  48 hours | 1.8 (0.5) | 1.3 (0.5)
  14 days | 1.4 (0.6) | 1.4 (0.8)
  30 days | 1.2 (0.6) | 1.3 (0.7)

9. Secondary Outcome: Number of Participants With Clinical Events
Time Frame: from randomization to second CMR
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Alfa | Placebo
Number analyzed (Participants) | 125 | 97
Participants
  Death | 1 | 0
  Recurrent myocardial infarction | 2 | 0
  Unstaged Percutaneous Coronary Intervention | 6 | 0
  Coronary Artery Bypass Graft | 0 | 1
  Stroke | 1 | 0
  Stent thrombosis | 3 | 0
  Left Ventricular thrombus | 3 | 2
  New or worsening Congestive Heart Failur | 5 | 2

ADVERSE EVENTS:
Groups:
- Epoetin Alfa: Patients who received active study medication
- Placebo: Patients who received placebo
Arm/Group | Epoetin Alfa | Placebo
Serious Adverse Events (participants affected / at risk) | 25/125 | 10/97
Other Adverse Events (participants affected / at risk) | 55/125 | 36/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epoetin Alfa (N=125) | Placebo (N=97)
Stent Thrombosis (Cardiac disorders) | 3 (3) | 0 (0) — Stent thrombosis was acute (7 hours after study medication) in one participants who received 60000 U dose of epoetin alka and subacute (5 days to 14 days)after receiving study medication
MI (Cardiac disorders) | 2 (2) | 0 (0) — Recurrent MI as a result of stent thrombosis
Renal Failure (Renal and urinary disorders) | 1 (1) | 2 (2) — 90y male 15000 U developed renal failure and subsequently died of heart failure 2 weeks after enrollment
Stroke (Cardiac disorders) | 1 (1) | 0 (0)
Death (Cardiac disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 2
Coronary disease (Cardiac disorders) | 0 | 1
Dressler's syndrome (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 3 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Heparin-induced thrombocytopenia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 4 | 1
Pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa (N=125) | Placebo (N=97)
Cardiac disorders (Cardiac disorders) | 26 | 13
Gastrointestinal disorders (Gastrointestinal disorders) | 12 | 6
General disorders and administration site conditions (General disorders) | 15 | 12
Investigations (Investigations) | 9 | 8
Psychiatric disorders (Psychiatric disorders) | 10 | 1
Vascular disorders (Vascular disorders) | 9 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less